CLINICAL TRIAL: NCT02175407
Title: A Phase 1, One Sequence, Cross-over Pharmacokinetic Study to Assess the Interaction Between ASP1707 and Itraconazole, a CYP3A and P-gp Inhibitor in Healthy Female Subjects
Brief Title: A Study to Assess the Interaction Between ASP1707 and Itraconazole in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1707-CL-0030; 2013-005370-21 (EudraCT Number)
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Pharmacokinetics; DDI (Drug-Drug Interaction); Healthy Subjects
Keywords: Healthy subjects; ASP1707; Itraconazole
MeSH Terms: interventions — opigolix; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP1707 alone (Experimental)
  Interventions: Drug: ASP1707
- ASP1707 + itraconazole (Experimental)
  Interventions: Drug: ASP1707; Drug: itraconazole

INTERVENTIONS:
Drug: ASP1707 — oral
Drug: itraconazole — oral
  Arms: ASP1707 + itraconazole

SUMMARY:
The purpose of this study to explore the effect of multiple oral doses of itraconazole on the pharmacokinetics of a single oral dose of ASP1707 in healthy female subjects. This study will also evaluate the safety and tolerability of a single oral dose of ASP1707 alone and in combination with itraconazole.

DETAILED DESCRIPTION:
Subjects will be confined in the clinical unit for up to 15 days.

ELIGIBILITY:
Inclusion Criteria:

* Female subject must be either of non child bearing potential, post-menopausal prior to screening, or documented surgically sterile. Or, if of childbearing potential, must agree not to try to become pregnant during the study and for 28 days after the final study drug administration, must have a negative urine pregnancy test at Day -1 and, if heterosexually active, agree to consistently use two forms of highly effective form of birth control starting at screening and throughout the study period and for 28 days after the final study drug administration.
* Female subject must not be breastfeeding at screening or during the study period, and for 28 days after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the study period, and for 28 days after the final study drug administration.

Exclusion Criteria:

* Female subject who has been pregnant within 6 months prior to screening assessment or breast feeding within 3 months prior to screening.
* Subject uses grapefruit (more than 3x 200 mL) or marmalade (more than three times) in the week prior to admission to the Clinical Unit until ESV, as reported by the subject.
* Subject is a vulnerable subject (e.g., subject kept in detention).

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of ASP1707 (=R-enantiomer), AS1948006 and the sum of ASP1707 and AS1948006 with itraconazole: AUCinf | Day 1-15
  Area under the plasma concentration - time curve from time zero to infinity (AUCinf)
Pharmacokinetic parameter of ASP1707 (=R-enantiomer), AS1948006 and the sum of ASP1707 and AS1948006 without itraconazole: AUCinf | Day 1-15
Pharmacokinetic parameter of ASP1707 (=R-enantiomer), AS1948006 and the sum of ASP1707 and AS1948006 with itraconazole: Cmax | Day 1-15
  Maximum concentration (Cmax)
Pharmacokinetic parameter of ASP1707 (=R-enantiomer), AS1948006 and the sum of ASP1707 and AS1948006 without itraconazole: Cmax | Day 1-15

SECONDARY OUTCOMES:
Composite of pharmacokinetics of ASP1707 (=R-enantiomer), AS1948006 and the sum of ASP1707 and AS1948006 concentration with itraconazole: AUClast, tmax, t1/2, AUCinf (%extrap), tlag, MRT, λz, CL/F, Vz/F, TER and MPR | Day 1-15
  Area under the plasma concentration - time curve from time zero to time of last measurable concentration (AUClast), Time to attain Cmax (tmax), apparent terminal elimination half life (t1/2), area under the concentration-time curve from the time of dosing extrapolated to time infinity (AUCinf [%extrap]), absorption lag time (tlag), Mean Residence Time (MRT), terminal elimination rate constant (λz), apparent total systemic clearance (CL/F) (ASP1707 (=R-enantiomer) only), apparent volume of distribution during terminal elimination phase (Vz/F) (ASP1707 only), total exposure ratio (TER) and metabolite-parent ratio (MPR) (AS1948006 only)
Composite of pharmacokinetics of ASP1707 (=R-enantiomer), AS1948006 and the sum of ASP1707 and AS1948006 concentration without itraconazole: AUClast, tmax, t1/2, AUCinf (%extrap), tlag, MRT, λz, CL/F, Vz/F, TER and MPR | Day 1-15
  CL/F (ASP1707 (=R-enantiomer) only), Vz/F (ASP1707 only), MPR (AS1948006 only)
Composite of pharmacokinetics of itraconazole and hydroxy itraconazole concentrations with ASP1707 (=R-enantiomer), AS1948006 and the sum of ASP1707 and AS1948006: AUCtau, tmax, Cmax, MPR (hydroxy itraconazole only), Ctrough | Days 4-15
  Area under the plasma concentration - time curve between consecutive dosing (AUCtau), plasma concentration at the end of a dosing interval at steady state (Ctrough)

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Lead, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- PAREXEL International GmbH, Berlin, Germany